CLINICAL TRIAL: NCT02218359
Title: A Randomized Double-Blind, Placebo-Controlled, Crossover to Open Label, Phase 2 Study of Aerosolized Amikacin and Fosfomycin Delivered Via the Investigational eFlow® AFIS Inline System in Mechanically Ventilated Patients With Gram-negative and/or Gram-positive Bacterial Colonization
Brief Title: Aerosolized Amikacin and Fosfomycin in Mechanically Ventilated Patients With Gram-negative and / or Gram-positive Bacterial Colonization
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Cardeas Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CAP-01-103
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Pneumonia, Bacterial
Keywords: Gram-negative pneumonia; Aerosol antibiotics; Mechanical ventilation; Amikacin; Fosfomycin; Pneumonia, Bacterial; Pneumonia; Bacterial Infections; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Anti-Bacterial Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; MRSA
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia; Bacterial Infections; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amikacin Fosfomycin Inhalation Solution (Experimental): 300 mg of amikacin and 120 mg of fosfomycin to be administered by aerosol via the AFIS Inline System.
  Interventions: Drug: Amikacin Fosfomycin Inhalation Solution
- Aerosolized Placebo (Placebo Comparator): Aerosolized placebo to be administered by aerosol using the AFIS Inline System.
  Interventions: Drug: Aerosolized placebo; Drug: Amikacin Fosfomycin Inhalation Solution

INTERVENTIONS:
Drug: Amikacin Fosfomycin Inhalation Solution — 300 mg of amikacin and 120 mg of fosfomycin twice daily for 10 days to be administered by aerosol via the AFIS Inline System
  Other Names: Amikacin Fosfomycin Inhalation System (AFIS); eFlow Inline System
  Arms: Amikacin Fosfomycin Inhalation Solution
Drug: Aerosolized placebo — Placebo twice daily for Days 1 -5 to be administered by aerosol using the eFlow Inline System.
  Other Names: eFlow Inline System
  Arms: Aerosolized Placebo
Drug: Amikacin Fosfomycin Inhalation Solution — Open-label crossover for all patients Days 6-10
  Other Names: Amikacin Fosfomycin Inhalation System (AFIS); eFlow Inline System

SUMMARY:
To demonstrate the safety and efficacy of adjunctive therapy with the Amikacin Fosfomycin Inhalation System (AFIS) versus aerosolized placebo in mechanically ventilated patients with Gram-negative and / or Gram-positive bacterial colonization.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate the safety and efficacy of the amikacin fosfomycin inhalation system (AFIS). AFIS consists of amikacin solution (AMS) and fosfomycin solution (FFS), delivered by aerosol to the lungs via the Investigational eFlow AFIS Inline System (AFIS Inline System) with tamper evident reservoir. Patients will be randomized to receive 5 days of treatment with either AFIS or placebo, followed by all patients receiving open label AFIS for five days. The primary efficacy endpoint is the change from baseline in tracheal aspirate Gram-negative and/or Gram-positive bacterial density at the end of the 5-day randomized course of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females, ≥ 18 years and ≤ 80 years of age
* Intubated and mechanically-ventilated
* Presence of Gram-negative and/or Gram-positive organism(s) by culture of respiratory secretions from a sample obtained within the previous 7 days

Exclusion Criteria:

* History of hypersensitivity to amikacin or fosfomycin.
* Diagnosis of pneumonia, defined as presence of a new or progressive infiltrate(s) on chest radiograph (within 7 days prior to screening), as determined by the treating physician
* Use of systemic antibiotics with efficacy against likely respiratory tract pathogens at the time of randomization
* Severe acute respiratory distress syndrome (defined as PaO2/FiO2 ≤ 100 mmHg and diffuse infiltrates on Chest X-ray)
* Refractory septic shock (severe sepsis plus unstable hypotension, in spite of adequate fluid resuscitation and vasopressors)
* Evidence of significant renal impairment (serum creatinine > 4.0 mg/dL within 24 hours prior to screening) . If serum creatinine is > 2.0 mg/dL, site must be capable of performing continuous renal replacement therapy, if clinically indicated. Patients with serum creatinine > 4.0 mg/dL and being treated with continuous renal replacement therapy (continuous venous-venous hemofiltration or continuous venous-venous hemodialysis) or chronic hemodialysis are eligible
* Evidence of ototoxicity (history of hearing aid use prior to current hospitalization)
* Evidence of hepatotoxicity (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3X the upper limit of normal value within 24 hours prior to screening)
* Any of the following conditions that interfere with the assessment or interpretation of the diagnosis or response to therapy: chest trauma with loss of stability of the thoracic cage following a fracture of the sternum, ribs, or both; increased amounts of fluid in the lung cavities requiring chest tube drainage; lung cancer within the last 2 years; lung abscess(s); anatomical bronchial obstruction; suspected atypical pneumonia; chemical pneumonitis (e.g., inhalation injury); cystic fibrosis; congestive heart failure (leading to a PaO2/FiO2 ratio ≤ 100 mmHg and diffuse infiltrates on Chest X-ray)
* Immunocompromised patients, including those with neutropenia NOT due to the current infection (absolute neutrophil count < 500/mm³), leukemia, lymphoma, human immunodeficiency virus (HIV) infection with CD4 count < 200 cells/mm3, or splenectomy; those who are early post-transplantation, are on cytotoxic chemotherapy, or are on high-dose steroids (e.g., > 40 mg of prednisone or its equivalent [> 160 mg hydrocortisone, > 32 mg methylprednisolone, > 6 mg dexamethasone, > 200 mg cortisone] daily for > 2 weeks)
* Positive urine and/or serum beta-hCG pregnancy test (only in women of reproductive age)
* Participating in or has participated in other investigational interventional studies (drug or device) within the last 30 days (or 5 times the half-life of the previously administered investigational compound, whichever is longer) prior to study treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in tracheal aspirate Gram-negative and Gram-positive bacterial density | 5 day randomized course of study drug
  Change from baseline in tracheal aspirate Gram-negative and Gram-positive bacterial density at the end of the 5-day randomized course of study drug

SECONDARY OUTCOMES:
Microbiological response rate in patients with multidrug resistant Gram-negative bacteria | Day 5
  Microbiological response rates at Day 5 in patients whose pre-study treatment tracheal aspirate culture was positive for multidrug resistant (MDR) Gram-negative bacteria
Eradication of bacteria | Days 10, 21, and 28
  Eradication of bacteria at Days 10, 21, and 28
Clinical worsening | Day 1 - Day 28
  Clinical worsening (defined as requiring institution of IV antibiotics) from Day 1 through Day 28
Microbiological response rates | Day 10
  Microbiological response rates at Day 10 in all patients
Microbiological response rates in patients with MRSA | Day 5
  Microbiological response rates at Day 5 in patients whose pre-study treatment tracheal aspirate culture was positive for methicillin resistant Staphylococcus aureus (MRSA)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, M.D., Study Director — Cardeas Pharma

REFERENCES:
- See also: MedlinePlus related topics: Antibiotics — http://www.nlm.nih.gov/medlineplus/antibiotics.html
- See also: MedlinePlus related topics: Pneumonia — http://www.nlm.nih.gov/medlineplus/pneumonia.html
- See also: Drug Information available for amikacin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0037517285&QV1=AMIKACIN
- See also: Drug information available for fosfomycin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0023155024&QV1=FOSFOMYCIN
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks